CLINICAL TRIAL: NCT06524843
Title: Generation of Synthetic Patient Data (RAW) for Risk Evaluation of Bone Metastases Derived From Carcinoma
Brief Title: Fracture Risk Evaluation of Bone Metastases Derived From Carcinoma
Status: Recruiting | Type: Observational
Sponsor: Costantino Errani (Other)
Responsible Party: Sponsor-Investigator, Costantino Errani, MD, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: FRAIL-RAW
Record Dates: First submitted 2024-07-23; First posted 2024-07-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Bone Metastases
Keywords: Bone metastases; Prediction model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Male and female patients affected by bone metastases derived from carcinoma, treated at Rizzoli Orthopaedic Institute from 01/01/2010 to 31/12/2022
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — Analysis and review of imaging and clinical data

SUMMARY:
From the archives of the Rizzoli institute all patients (approximately 750) treated for bone metastases from 01/01/2010 to 31/12/2022.

A review will be made from the medical records, radiological imaging, and histological data of these patients

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of bone metastasis from carcinoma, regardless of the type of carcinoma, and of the number and location of the metastases
* Availability of imaging and clinical data
* Availability of at least one follow-up during the last 12 months form diagnosis

Exclusion Criteria:

* At least one inclusion creteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female adult patients, affected by bone metastases derived from carcinoma, treated at Rizzoli Ortopaedic institute from 01/01/2010 to 31/12/2022.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Creation a dataset of clinical data and diagnostic images | At baseline (Day 0)
  Creation a dataset of clinical data and diagnostic images, called RAW, relating to patients suffering from metastatic bone cancer that will be used by the unit UNICH to create innovative models for fracture risk prediction and of life expectancy based on various patient clinical parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mirels H. Metastatic disease in long bones: A proposed scoring system for diagnosing impending pathologic fractures. 1989. Clin Orthop Relat Res. 2003 Oct;(415 Suppl):S4-13. doi: 10.1097/01.blo.0000093045.56370.dd. PMID 14600587
- [Background] Coleman RE. Clinical features of metastatic bone disease and risk of skeletal morbidity. Clin Cancer Res. 2006 Oct 15;12(20 Pt 2):6243s-6249s. doi: 10.1158/1078-0432.CCR-06-0931. PMID 17062708